CLINICAL TRIAL: NCT02431533
Title: The Efficacy of PX0612 In The Treatment Of Irritable Bowel Syndrome: A Randomized, Double-Blind Placebo Controlled Clinical Trial
Brief Title: The Efficacy of PX0612 In The Treatment Of Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmabiotix Inc (Industry)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-PBI-2012
Record Dates: First submitted 2015-04-09; First posted 2015-05-01 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS-D; diarrhea predominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic PX0612 (Experimental): PX0612 is a probiotic contained in a veggie capsule.
  Interventions: Dietary Supplement: PX0612
- Di-Calcium Phosphate (Placebo Comparator): Patients in the 'placebo' group will receive the placebo capsules. The main ingredient in the placebo capsule is Di-Calcium Phosphate
  Interventions: Dietary Supplement: Di-Calcium Phosphate

INTERVENTIONS:
Dietary Supplement: PX0612 — PX0612 is a probiotic contained in a veggie capsule.
  Arms: Probiotic PX0612
Dietary Supplement: Di-Calcium Phosphate — Patients in the 'placebo' group will receive the placebo capsules. The main ingredient in the placebo capsule is Di-Calcium Phosphate
  Arms: Di-Calcium Phosphate

SUMMARY:
IBS is a disorder of movement in the gut. People who have IBS may have diarrhea, constipation, or alternating bouts of both. IBS is not caused by injury or illness. Often the only way doctors can diagnose it is to rule out other conditions through testing.

DETAILED DESCRIPTION:
Probiotics, particularly Bifidobacterium infantis, Sacchromyces boulardii, Lactobacillus plantarum and combination probiotics may help regulate how often people with IBS have bowel movements. Probiotics may also help relieve bloating from gas. Research is continuing to determine which probiotics are best to treat IBS.

PX0612

PX0612 is a probiotic which is composed of the following ingredients contained in a veggie capsule, being one dose:

Bacillus coagulans 200 million colony forming units 16.0mg Bacillus subtilis 100 million colony forming units 4.8mg Enterococcus faecium 100 million colony forming units 0.6mg Fructo-oligosacharride a nutrient for the packaged product 600.0mg Total 621.4 mg Bacillus coagulans is a non-pathogenic, Gram positive, spore forming bacteria that produces lactic acid. Though not normally found in the gut. Bacillus coagulans strains have been used as general nutritional supplements and agents to control constipation and diarrhea in humans and animals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 - 65 years old
* Signed informed consent
* Mild to moderate (using Functional Bowel Disorder Severity Index (FBDSI)) IBS-Diarrhea patient:

  * IBS definition will be based on Rome criteria;

The symptoms of IBS must persist for at least 3 months and must include:

1. Abdominal pain or discomfort which is relieved by defecation, and/or associated with a change in frequency of stool and/or consistency of stool
2. At least two of the following, at least a quarter of occasions or days (25%):

A. Altered stool frequency (> 3 bowel movements/day or < 3 bowel movements/week) B. Altered stool form (lumpy/hard or loose/watery stools) C. Altered stool passage (straining, urgency or feeling of incomplete evacuation) D. Passage of mucus E. Bloating or feeling of abdominal distention

Note: Diarrhea is defined as having loose watery stools at least three times per day

Exclusion Criteria:

* The patient will be excluded from the study if:

  * Assessment by the treating investigator showed an evidence for cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematologic/immunologic, head, ears, eyes, nose and throat, dermatologic/psychiatric, allergy, major surgery or other diseases as revealed by history, physical examination and existing laboratory assessments which may interfere with the administration or 5 | P a g e

PX0612 In The Treatment Of Irritable Bowel Syndrome:

assessment of study medication. This should be confirmed by a pre-study medical examination performed 2 weeks prior the study.

* Pregnant or lactating
* Females at child bearing age will be excluded unless they are using acceptable birth control measures (i.e. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence or a vasectomized partner)
* Patients requiring treatments with non-permitted medication (i.e. 5-HT3 antagonist, spasmolytics, anticholinergics, cholestyramine, anti flatulence agents, metoclopramide, gastric-anti secretory agents (proton pump inhibitors; for indications other than Gastroesophageal Reflux Disease (GERD)), narcotics, anti-diarrheal drugs, and systemic steroids)
* Patients requiring the use of antibiotics either in medicine form of natural (e.g. grapefruit seed extract, olive leaf extract, oil of oregano, colloidal silver and highly concentrated garlic preparations)
* Exercise and the use of complementary and alternative medicine for IBS symptoms (i.e. peppermint oil, cognitive behavior therapy) during the study should be maintained at the same level prior to the study.
* Patients exceeding the treatment limits of permitted medication [(more than 2 days/week during the study period): alginate, antacids and analgesics (limited to acetaminophen ≤ 1000 mg/day, acetylsalicylic acid or NSAIDS no more than 2 tablets/day), (stable dose throughout the study period, anti-depressants (must be on a stable dose > 3 months), fiber supplements, psyllium hydrophilic mucilloid, gastric anti secretory agents (only for GERD patients who are on a stable dose > 3 months; patients should be able to differentiate between IBS and GERD symptoms), acetylsalicylic acid ≤ 325 mg/day, sedatives. Deliverance medications: Mild laxatives only if necessary.]. Any other medications can be used without limits based on the clinical judgment of the treating investigator.
* Being in another clinical trial 4 weeks before entering the study
* Constipated IBS patients
* IBS-Diarrhea patients with un-treated lactose intolerance
* Regular use of probiotics or using other probiotics during the course of the study
* Patients allergic to milk or soy products
* Patients using catheters
* Patients presented with rectal bleeding, weight loss, iron deficiency anemia, nocturnal symptoms and a family history of colorectal cancer, inflammatory bowel disease and celiac spruce
* Patients over 50 diagnosed with Irritable Bowel Syndrome who have not had a colonoscopy in the last 5 years
* Patients who have allergies for the active ingredients or any of the exepients
* Patients presented with any immune-compromised condition (such as AIDS, lymphoma, long term corticosteroid treatment)
* Patients presented with nausea, vomiting and fever 6 |

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Richer, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Longstreth GF, Wilson A, Knight K, Wong J, Chiou CF, Barghout V, Frech F, Ofman JJ. Irritable bowel syndrome, health care use, and costs: a U.S. managed care perspective. Am J Gastroenterol. 2003 Mar;98(3):600-7. doi: 10.1111/j.1572-0241.2003.07296.x. PMID 12650794
- [Background] Drossman DA. Review article: an integrated approach to the irritable bowel syndrome. Aliment Pharmacol Ther. 1999 May;13 Suppl 2:3-14. doi: 10.1046/j.1365-2036.1999.0130s2003.x. PMID 10429736
- [Background] Schoenfeld P, Talley NJ. Measuring successful treatment of irritable bowel syndrome: is "satisfactory relief " enough? Am J Gastroenterol. 2006 May;101(5):1066-8. doi: 10.1111/j.1572-0241.2006.00519.x. PMID 16696786
- [Background] Dolin BJ. Effects of a proprietary Bacillus coagulans preparation on symptoms of diarrhea-predominant irritable bowel syndrome. Methods Find Exp Clin Pharmacol. 2009 Dec;31(10):655-9. doi: 10.1358/mf.2009.31.10.1441078. PMID 20140275

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Started | 25 | 25
Completed | 23 | 22
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Developed Exclusionary criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Count of Participants; unit: Participants]
  >18 and <65 years of age | 25 | 25 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Bowel Movements Per Day [Mean (Full Range); unit: bowel movements/day] — Frequency of Bowel Movements Per Day, measured as total number of bowel movements per day.
  bowel movements/day | 2.35 [1.96 to 2.73] | 2.39 [1.87 to 2.73] | 2.37 [1.87 to 2.73]
Functional Bowel Disorder Severity Index [Mean (Full Range); unit: units on a scale] — , higher score= greater severity total score range from 0-500
  units on a scale | 272 [243 to 301] | 234 [196 to 271] | 253 [196 to 301]
Abdominal Pain- higher the number, greater the pain [Mean (Full Range); unit: units on a scale] — The scale of pain ranges from 0-4, 4 indicating incapacitating pain.
  units on a scale | 1.34 [1.13 to 1.55] | 1.2 [1.03 to 1.38] | 1.27 [1.03 to 1.55]
Stool Consistency [Mean (Full Range); unit: units on a scale] — 1= solid stools 7= loose stools diarrhea
  units on a scale | 5.08 [1 to 7] | 4.73 [1 to 7] | 4.91 [1 to 7]
Short Form 36 Health Survey [Mean (Standard Deviation); unit: units on a scale] — Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. Scoring is based on software program.
  units on a scale | 48.92 (7.38) | 50.49 (7.44) | 49.71 (7.41)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Bowel Movements (Stool Frequency) Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period.
Description: For each patient stool frequency was measured as a number of bowel movements per day. To compare stool frequency before and after the treatment, the average for the first 2 run-in weeks (day 1 - day 14) and the last 2 weeks (day 78 - day 91) was calculated.
  A higher mean score indicates a better outcome, a greater reduction in bowel movements/day and is a positive change.
  Placebo group- min: -.43 max: 1.43
  Study group- min: -.43 max: 1.50
Time Frame: Baseline (days 1-14) compared to Weeks 10 and 11 of treatment (days 78-91)
Population: The total number of participants analyzed for Di-Calcium Phosphate differs from the overall analysis number as the data for one of these participants was not sufficient for use (not enough data available to evaluate) for this particular outcome.
Measure: Mean (95% Confidence Interval); unit: bowel movements/day
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 21
bowel movements/day | .46 [.25 to .67] | .21 [-.04 to .46]

2. Secondary Outcome: Differences in Upper Gastrointestinal Symptoms Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period.
Description: Mean change in heartburn between baseline (days 1-14) and weeks 10 and 11 (days 78-91) between the two groups.
  A higher mean value indicates a greater reduction in heartburn, better outcome.
  Analog Scale from 0-4 was used by participants to rate upper GI symptoms of heartburn (0= no heartburn, 4= incapacitating).
  Placebo group- Min: -2.00 Max: 3.00
  Treatment group- Min: -2.00 Max: 2.00
Time Frame: Baseline (days 1-14) compared to Weeks 10 and 11 of treatment (days 78-91)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | .09 [-.30 to 0.48] | -.09 [-.48 to .29]

3. Secondary Outcome: Differences in Upper Gastrointestinal Symptoms- Vomiting Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period.
Description: vomit scale used was from 0-4, the higher the number, the worse the outcome Mean change in vomiting between baseline and week 12 between the two groups. A higher mean value indicates a greater reduction in vomiting, better outcome.
  Analog Scale from 0-4 was used by participants to rate upper GI symptoms of vomiting(0= none, 4= incapacitating).
  Placebo group- Min: 0 Max: 0
  Treatment group- Min: -3.00 Max: 0
Time Frame: Baseline compared to Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | -.22 [-.51 to .07] | 0 [0 to 0]

4. Secondary Outcome: Changes in the Patient's Assessment of Their Quality of Life Using Short Form(SF)-36 Health Survey PCS (Physical Component Score)
Description: Differences in quality of life phusical component score using SF-36 between the 'intervention' group and the 'placebo' group over the study period. Baseline PCS scores were compared to the end of the study time point. The mean difference between the 2 time points was measured.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. Scoring is based on software program.
  Placebo group- Min: -16.16 Max: 6.25
  Treatment group- Min: -16.42 Max: 5.46
  The total number of participants analyzed in each group differs as a result of the number of participants that either withdrew or were withdrawn in the study. Data were analyzed and compared for participants that completed the study.
Time Frame: Baseline compared to Week 12 (end of study)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 21
units on a scale | -2.27 [-4.35 to -.19] | -2.05 [-4.53 to .43]

5. Secondary Outcome: Differences in Abdominal Pain/Discomfort Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period.
Description: Outcome measure is the mean change of abdominal pain, on a scale of 0-4 (0= no pain, 4= incapacitating pain), between baseline and Weeks 10 and 11. A larger change in average abdominal pain indicates a greater reduction in mean abdominal pain score, better outcome.
  Min=-.067 for treatment group Min= -.99 for placebo group Max= 1.14 for treatment group Max= 1.63 for placebo group The total number of participants analyzed in each group differs as a result of the number of participants that either withdrew or were withdrawn in the study. Data were analyzed and compared for participants that completed the study.
Time Frame: Baseline (days 1-14) compared to Weeks 10 and 11 of treatment (days 78-92)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 21
units on a scale | 0.35 [0.13 to 0.56] | 0.44 [0.16 to 0.72]

6. Secondary Outcome: Differences in Stool Consistency Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period.
Description: The stool consistency before and after the treatment was compared, the average for the first 2 run-in weeks (day 1 - day 14) and the last 2 weeks (day 78 - day 91) was calculated. A higher mean outcome indicates a greater reduction in loose stool/diarrhea (better outcome).
  Bristol Stool Chart (1=severe constipation to 7 =severe diarrhea) was the scale used for measurement. The participant reported outcomes were averaged at above time points for comparison.
  Min for placebo group: -.70 Max for treatment group: 2.57 Max for placebo group: 1.88
  The total number of participants analyzed in each group differs as a result of the number of participants that either withdrew or were withdrawn in the study. Data were analyzed and compared for participants that completed the study.
Time Frame: Baseline (days 1-14) compared to Weeks 10 and 11 of treatment (days 78-92)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 21
units on a scale | 0.51 [0.16 to 0.86] | 0.46 [0.14 to 0.78]

7. Secondary Outcome: Differences in Stool Frequency Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period.
Description: Number of stools/day
Time Frame: Baseline (days 1-14) compared to Weeks 10 and 11 of treatment (days 78-92)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: stools/day
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 21
stools/day | 2.35 [1.96 to 2.73] | 2.39 [1.87 to 2.73]

8. Secondary Outcome: Differences in Upper Gastrointestinal Symptoms- Early Satiety
Description: Differences Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period. Change in rate of early satiety on a scale from 0-4 (higher the score, the worse the outcome) Mean change in early satiety between baseline and week 12 between the two groups.
  A higher mean value indicates a greater reduction in early satiety, better outcome.
  Analog Scale from 0-4 was used by participants to rate upper GI symptoms of early satiety (0= none, 4= incapacitating).
  Placebo group- Min: -2.00 Max: 1.00
  Treatment group- Min: -2.00 Max: 2.00
Time Frame: Baseline compared to Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | .26 [-.13 to .66] | -.27 [-.66 to .12]

9. Secondary Outcome: The Difference in Change of Postprandial Fullness Severity
Description: Differences Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period. Mean change in postprandial fullness between baseline and week 12 between the two groups.
  A higher mean value indicates a greater reduction in a postprandial fullness, better outcome.
  Analog Scale from 0-4 was used by participants to rate upper GI symptoms of postprandial fullness (0= no postprandial fullness, 4= incapacitating postprandial fullness).
  Placebo group- Min: -1.00 Max: 2.00
  Treatment group- Min: -1.00 Max: 2.00
Time Frame: Baseline compared to Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | .22 [-.10 to .54] | .18 [-.22 to .58]

10. Secondary Outcome: Upper Gastrointestinal Symptoms of Prolonged Digestion
Description: Differences Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period. Mean change in prolonged digestion between baseline and week 12 between the two groups.
  A higher mean value indicates a greater reduction in prolonged digestion, better outcome.
  Analog Scale from 0-4 was used by participants to rate upper GI symptoms of prolonged digestion (0= none, 4= incapacitating).
  Placebo group- Min: -2.00 Max: 1.00
  Treatment group- Min: -1.00 Max: 3.00
Time Frame: Baseline compared to Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | .35 [-.03 to .73] | -.05 [-.42 to .33]

11. Secondary Outcome: Upper Gastrointestinal Symptom of Nausea
Description: Differences Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period. Mean change in nausea between baseline and week 12 between the two groups.
  A higher mean value indicates a greater reduction in nausea, better outcome.
  Analog Scale from 0-4 was used by participants to rate upper GI symptoms of nausea(0= none, 4= incapacitating).
  Placebo group- Min: 0.00 Max: 2.00
  Treatment group- Min: -1.00 Max: 1.00
Time Frame: Baseline and Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | .09 [-.2 to .38] | .32 [.03 to .6]

12. Secondary Outcome: FBDSI (Functional Bowel Disease Severity Index)
Description: Differences Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period. Mean change in FBDSI score between baseline and week 12 between the two groups.
  A higher mean value indicates a greater reduction in bowel disease severity, better outcome.
  Functional Bowel Disease Severity Index was the scale used to determine this outcome. The range on this scale is from 0-500, with 500 indicating the most severe functional bowel disease.
  Placebo group- Min: -10.00 Max: 350.00
  Treatment group- Min: 0 Max: 300.00
Time Frame: Baseline compared to Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
units on a scale | 96.26 [66.04 to 126.48] | 133.41 [93.22 to 173.60]

13. Post Hoc Outcome: Participants With 30% or More Reduction in Functional Bowel Disease Severity Index (FBDSI)
Description: Differences Between the 'Intervention' Group and the 'Placebo' Group Over the Study Period. Mean change in FBDSI score between baseline and week 12 between the two groups.
  A higher mean value indicates a greater reduction in bowel disease severity, better outcome.
  Functional Bowel Disease Severity Index was the scale used to determine this outcome. The range on this scale is from 0-500, with 500 indicating the most severe functional bowel disease.
  This measure represents the total number of participants that had a 30% or greater reduction in FBDSI score.
Time Frame: Baseline assessment compared to visit 5 assessment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
Participants | 10 | 3

14. Post Hoc Outcome: Unplanned Analysis- Participants With 30% or Greater Reduction in Stool Frequency/Day
Description: Percentage of participants with a greater than 30% reduction in the number of stools/day.
Time Frame: Baseline (days 1-14) compared to Weeks 10 and 11 of treatment (days 78-91)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
Number analyzed (Participants) | 23 | 22
percentage of participants | 35 [18 to 56] | 9 [2.1 to 31]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during study participation over a 14 week period for each participant.
Description: Reporting was performed as per GCP standards
Arm/Group | Probiotic PX0612 | Di-Calcium Phosphate
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 7/25 | 15/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic PX0612 (N=25) | Di-Calcium Phosphate (N=25)
Heartburn (Gastrointestinal disorders) | 3 (3) | 1 (1)
increased bloating/gas (Gastrointestinal disorders) | 1 (3) | 2 (3)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased Restless Leg Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Lower back pain (General disorders) | 0 (0) | 2 (2)
Migraine/headache (General disorders) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight gain (General disorders) | 0 (0) | 1 (1)
Ear pain/dizziness (General disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Statistical Analysis (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02431533/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Final Report Version (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT02431533/SAP_001.pdf